CLINICAL TRIAL: NCT01091233
Title: The Influence of Paracentesis on Intra-abdominal Pressure and Kidney Function in Critically Ill Patients With Liver Cirrhosis and Ascites: an Observational Study
Status: Withdrawn | Type: Observational
Why Stopped: logistical problems
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Other Study IDs: 2009/722
Record Dates: First submitted 2010-03-19; First posted 2010-03-23 (Estimated); Last update posted 2021-07-08 (Actual); Status verified 2021-07

CONDITIONS: Critically Ill; Liver Cirrhosis; Ascites
Keywords: Critically ill patients; liver cirrhosis; ascites requiring Paracentesis
MeSH Terms: conditions — Critical Illness; Liver Cirrhosis; Ascites | interventions — Paracentesis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Paracentesis: Paracentesis as indicated according to the treating physician (the indication for Paracentesis is not the subject of study)
  Interventions: Procedure: paracentesis

INTERVENTIONS:
Procedure: paracentesis — as indicated according to the treating physician (the indication for Paracentesis is not the subject of study)

SUMMARY:
Patients with liver cirrhosis are at risk for development of renal failure, usually after a precipitating event such as infection or bleeding. This form of renal failure has a high morbidity and mortality and may be partly caused by increased intra-abdominal pressure secondary to ascites. Recent studies have shown that paracentesis (and the resulting decreased IAP) can increase urinary output and decrease renal arterial resistive index in patients with hepatorenal syndrome (a very pronounced form of renal failure in cirrhosis patients). The aim of this study is to evaluate the influence of Paracentesis on intra-abdominal pressure and kidney function in critically ill patients with liver cirrhosis and ascites across a wider range of kidney function. Kidney function will be evaluated using several estimates of glomerular filtration rate and measures of kidney injury i.e. cystatin C, serum NGAL, creatinine clearance, urinary output and renal arterial resistive index.

ELIGIBILITY:
Inclusion criteria:

* >18 y old
* Admitted to the ICU
* Known liver cirrhosis with ascites on clinical examination and/or ultrasound
* Sedated and mechanically ventilated
* Paracentesis deemed necessary by treating physician
* Arterial and central venous catheter in place
* Urinary catheter in place

Exclusion criteria:

* Previous inclusion in the same study
* Renal replacement therapy in place
* Urinary catheter contra-indicated
* Use of radiocontrast media within 72h before paracentesis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Critically ill patients with liver cirrhosis and ascites requiring Paracentesis according to treating physician
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2010-03; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Intra-abdominal pressure and kidney function before, during, immediately after and 12-24h after Paracentesis | 24h after paracentesis
  Kidney function parameters include 2h creatinine clearance, serum and urine creatinine, renal artery resistive index (measured via color Doppler), urinary output, serum cystatine C and NGAL measurement.

SECONDARY OUTCOMES:
The association between the change in IAP and kidney function | 24h after paracentesis
The relationship between the amount of fluid drained and any effect on IAP and kidney function | 24h after paracentesis
Cystatin C, NGAL, creatinine clearance, serum creatinine, urinary output and RI as measures of kidney injury in patients with liver cirrhosis and ascites | 24h after paracentesis

CONTACTS AND LOCATIONS:
Overall Officials: Eric Hoste, MD, PhD, Principal Investigator — University Hospital, Ghent
Locations (1):
- University Hospital Ghent, Ghent, Belgium

REFERENCES:
- See also: website University Hospital Ghent — http://www.uzgent.be